CLINICAL TRIAL: NCT02160184
Title: Nocturnal Insulin-Glucose in Hospital: Tight Control
Acronym: NIGHT CONTROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Mercedes Rigla, MD, PhD, Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: NIGHT CONTROL
Record Dates: First submitted 2014-06-09; First posted 2014-06-10 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2014-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (1):
- experimental (Experimental): Night under closed loop system
  Interventions: Device: Artificial pancreas system consisting of a predictive rule-based algorithm integrated on the Medtronic Portable Glucose Control System (PGCS)

INTERVENTIONS:
Device: Artificial pancreas system consisting of a predictive rule-based algorithm integrated on the Medtronic Portable Glucose Control System (PGCS)

SUMMARY:
The aim of the study is to assess the efficacy and safety of a closed-loop system consisting of a predictive rule-based algorithm integrated on the Medtronic Portable Glucose Control System (PGCS) in patients with type 1 diabetes for controlling the nocturnal and post-breakfast periods. Intervention will be to apply the automated closed-loop system by administering a subcutaneous insulin microbolus every 5 minutes depending on reading from a continuous glucose measurement (CGM) system.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Diabetes duration > 3 years
* Continuous Subcutaneous Insulin Infusion (CSII) treatment for more than 1 year
* A1c 6-9%
* No ketoacidosis during the previous 12 months
* Glomerular Filtration Rate (GFR) > 60 ml/kg/min m2
* Willingness of participate and signed and dated written informed consent in accordance with Good Clinical Practice

Exclusion Criteria:

* Gastroparesis
* Hypoglycemia unawareness
* Uncorrected visual impairment
* Deafness
* BMI> 35 kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of time in target range (3.9-8.0 mmol/l) YSI glucose during the in clinic overnight visit. | During the closed-loop period for each patient: 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Rigla, MD, PhD, Principal Investigator — Parc Tauli University Hospital
Locations (1):
- Parc Tauli University Hospital, Sabadell, Barcelona, Spain